CLINICAL TRIAL: NCT00842478
Title: Effectiveness of Dental Brushing for Preventing Ventilator-Associated Pneumonia
Acronym: RASPALL
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Joan XXIII de Tarragona. (Other)
Responsible Party: Jordi Rello, Hospital Universitari Joan XXIII
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FIS 06/0060
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2009-02

CONDITIONS: Ventilator-Associated Pneumonia; Nosocomial Pneumonia; Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Healthcare-Associated Pneumonia; Pneumonia | interventions — Toothbrushing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Raspall (Experimental)
  Interventions: Procedure: Toothbrushing
- Control (No Intervention)

INTERVENTIONS:
Procedure: Toothbrushing
  Arms: Raspall

SUMMARY:
Poor oral hygiene is associated with respiratory pathogen colonization and secondary lung infection.The possible association between oral care and incidence of VAP, and the role of dental plaque, mouth and tracheal colonization have not been firmly established. The investigators' hypothesis was that improving oral care with electrical toothbrushing might be effective in reducing the incidence of VAP.

ELIGIBILITY:
Inclusion Criteria:

* Adult intubated patients
* Without evidence of pulmonary infection (randomized within 12h of intubation if they were expected to remain ventilated for longer than 48 hours)

Exclusion Criteria:

* Absence of dental pieces
* Current diagnosis of pneumonia or massive bronchoaspiration
* Tracheostomy (or expected within 48 hours)
* Chlorhexidine allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2005-05

PRIMARY OUTCOMES:
Ventilator-Associated Pneumonia (VAP) | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Rello, MD, PhD, Principal Investigator — Hospital Universitari Joan XXIII
Locations (1):
- ICU, Hospital Universitari Joan XXIII, Tarragona, Tarragona, Spain

REFERENCES:
- [Derived] Pobo A, Lisboa T, Rodriguez A, Sole R, Magret M, Trefler S, Gomez F, Rello J; RASPALL Study Investigators. A randomized trial of dental brushing for preventing ventilator-associated pneumonia. Chest. 2009 Aug;136(2):433-439. doi: 10.1378/chest.09-0706. Epub 2009 May 29. PMID 19482956